CLINICAL TRIAL: NCT03271034
Title: Effect of Weight Loss on Body Composition and Metabolic Function in Women With Lipedema
Acronym: Lipedema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Lipedema Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201702107
Record Dates: First submitted 2017-08-29; First posted 2017-09-01 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Lipedema; Metabolism
Keywords: Lipedema; Metabolism; Body Composition; Fat Distribution; Immunology
MeSH Terms: conditions — Lipedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lean women with Lipedema (Experimental): Body composition, adipose tissue biology, insulin sensitivity assessed before and after low-calorie diet therapy to achieve 5-10% weight loss.
  Interventions: Dietary Supplement: Weight loss
- Women with Obesity and Lipedema (Experimental): Body composition, adipose tissue biology, insulin sensitivity and immune function/inflammation assessed before and after low-calorie diet therapy to achieve 5-10% weight loss.
  Interventions: Dietary Supplement: Weight loss

INTERVENTIONS:
Dietary Supplement: Weight loss — Participants will lose weight by utilizing a low caloric diet and meeting with a study dietitian and/or behaviorist weekly for ~4 months.

SUMMARY:
Lipedema is a disorder characterized by massive, bilateral accumulation of fat below the waist and in the legs. Enlargement of the lower extremities is often accompanied by leg pain and accumulation of fluid. Little is known about the functional changes that lead to fat accumulation and pain in women with lipedema. The goals of this project are to conduct a comprehensive characterization of abdominal and femoral fat tissues in lean and obese women with lipedema and to evaluate the potential effect of diet-induced weight loss as a therapy.

Once enrolled in the study, the following tests will be conducted on lean women with lipedema: characterization of body composition (fat tissue distribution), insulin sensitivity (response to insulin) and adipose tissue biology. The following tests will be conducted on obese women with lipedema: characterization of body composition (fat tissue distribution), insulin sensitivity (response to insulin), adipose tissue biology, and immune system function/inflammation. As control groups, we will compare body composition and insulin sensitivity to: i) women with obesity without lipedema who are matched on age, body mass index, total body fat mass, and percent body weight as fat; and ii) women who were lean and healthy to serve as a normal comparator for the 2 groups with obesity. Participants in the 2 control groups will enroll in a different study at Washington University (IRB# 201512086) where the same procedures will be performed to assess body composition and insulin sensitivity.

A second aim of the study is to determine the effect of diet-induced weight loss on body composition, insulin sensitivity, and adipose tissue biology in women with lipedema. The results from this second aim of the study will provide important insights on the efficacy of diet therapy in managing lipedema.

DETAILED DESCRIPTION:
Once informed consent has been obtained, participants will complete a screening visit that will include a medical history, physical examination, pregnancy test (for women of childbearing potential), blood tests, urine drug test, an oral glucose tolerance test, resting electrocardiogram (ECG), and questionnaires.

Baseline testing will be performed over 2 visits requiring 1 inpatient overnight stay and will require approximately 30 hours in total to complete testing. Testing will include magnetic resonance imaging scans to determine thigh fat mass; abdominal (belly) fat mass and liver fat content; DXA scan to assess whole-body and leg fat mass; blood samples; hyperinsulinemic-euglycemic clamp procedure to assess insulin sensitivity; immune system function/inflammation (performed exclusively in people with obesity and lipedema and BMI-matched controls); and adipose tissue (fat) biopsies.

Once Baseline Testing is completed, participants will start 5-10% dietitian and/or behaviorist guided weight-loss for about 4 to 6 months.

Participant will keep a food diary and have weekly visits (in person or remote) with a study dietitian and/or behaviorist.

After weight loss, the testing completed during baseline will be repeated.

Study procedures:

1. Medical history & physical exam
2. Urine drug/pregnancy Test
3. Blood pressure, pulse, height, weight
4. Electrocardiogram (ECG)
5. Blood tests for routine lab analyses
6. Oral glucose tolerance test (OGTT)
7. Screening Questionnaires
8. Dual energy X-ray absorptiometry (DXA) scan to assess whole-body and leg fat mass
9. Magnetic Resonance Imaging (MRI) to determine the amount of fat in the liver, abdomen (belly), and thigh.
10. Metabolism study (hyperinsulinemic-euglycemic clamp procedure) to assess how well insulin works to control blood glucose (sugar) concentrations.
11. Abdominal (belly) and thigh fat biopsies (women with obesity only)
12. Immune function (performed in people with obesity and lipedema only).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Lipedema
* Lean women with lipedema (BMI >19.5 kg/m² and <26.0 kg/m²)
* Women with obesity and lipedema (BMI >30.0 kg/m² and <50.0 kg/m²)

Exclusion Criteria:

* Medical, surgical or biological menopause
* Previous bariatric surgery
* Diagnosis of Type 2 Diabetes
* HbA1C <5.7%
* Structured exercise >2 days/week for ≥35 minutes of intense exercise (e.g., jogging, activity that cause heavy breathing and sweating) or ≥150 minutes per week of structured exercise (e.g., brisk walking)
* Unstable weight (>4% change in weight during the last 2 months before entering the study)
* Significant organ system dysfunction (e.g., diabetes, severe pulmonary, kidney or cardiovascular disease)
* Cancer or cancer that has been in remission for <5 years
* Polycystic Ovary Syndrome
* Major psychiatric illness
* Conditions that render participant unable to complete all testing procedures (e.g., severe ambulatory impairments, limb amputations, or metal implants that interfere with imaging procedures; coagulation disorders)
* Use of medications that are known to affect the study outcome measures (e.g., steroids, non-statin lipid-lowering medications) or increase the risk of study procedures (e.g., anticoagulants) and that cannot be temporarily discontinued for this study
* Smoke cigarettes >10 cigarettes/week
* Consume >14 units of alcohol per week
* Pregnant or lactating women
* Persons who are not able to grant voluntary informed consent
* Persons who are unable or unwilling to follow the study protocol or who, for any reason, the research team considers not an appropriate candidate for this study, including non-compliance with screening appointments or study visits.

Ages: 18 Years to 68 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2025-03-24 (Actual)

PRIMARY OUTCOMES:
Change in thigh subcutaneous adipose tissue volume | Before and after 5-10% weight loss (3-4 months)
  Thigh subcutaneous adipose tissue volume assessed by magnetic resonance imaging.
Whole-body insulin sensitivity | Baseline testing
  Whole-body insulin sensitivity determined by using the hyperinsulinemic-euglycemic clamp procedure between women with obesity and women with obesity and lipedema.

SECONDARY OUTCOMES:
Thigh subcutaneous adipose tissue volume | Baseline testing
  Thigh subcutaneous adipose tissue volume assessed by magnetic resonance imaging in women with obesity and lipedema, women with obesity and lean women.
Change in whole-body insulin sensitivity | Before and after 5-10% weight loss (3-4 months)
  Whole-body insulin sensitivity determined by using the hyperinsulinemic-euglycemic clamp procedure.
Leg fat mass | Baseline testing
  Leg fat mass will be assessed by dual-energy x-ray absorptiometry (DXA) in women with obesity and lipedema, women with obesity and lean women.
Change in leg fat mass | Before and after 5-10% weight loss (3-4 months)
  Leg fat mass will be assessed by dual-energy x-ray absorptiometry (DXA).
Adipose tissue immune cells | Baseline testing
  Immune cell numbers in upper and lower body subcutaneous adipose tissue stromal vascular fraction content assessed by flow cytometry in women with obesity and lipedema only.
Change in adipose tissue immune cells | Before and after 5-10% weight loss (3-4 months)
  Immune cell numbers in upper and lower body subcutaneous adipose tissue stromal vascular fraction content assessed by flow cytometry.

OTHER OUTCOMES:
Adipose tissue transcriptomics | Baseline testing
  Gene expression in abdominal and thigh subcutaneous adipose tissue will be analyzed and compared by using RNA sequencing in women with lipedema.
Change in abdominal subcutaneous adipose tissue transcriptomics | Before and after 5-10% weight loss (3-4 months)
  Gene expression in abdominal subcutaneous adipose tissue will be analyzed by using RNA sequencing.
Change in thigh subcutaneous adipose tissue transcriptomics | Before and after 5-10% weight loss (3-4 months)
  Gene expression in thigh subcutaneous adipose tissue will be analyzed by using RNA sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Klein, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Adipose tissue RNA sequencing will be uploaded to Gene Expression Omnibus (GEO).
Time Frame: Before publication of manuscript containing RNA sequencing results
Access Criteria: RNA sequencing results will be publicly available.
URL: https://www.ncbi.nlm.nih.gov/geo/

REFERENCES:
- [Result] Cifarelli V, Smith GI, Gonzalez-Nieves S, Samovski D, Palacios HH, Yoshino J, Stein RI, Fuchs A, Wright TF, Klein S. Adipose Tissue Biology and Effect of Weight Loss in Women With Lipedema. Diabetes. 2025 Mar 1;74(3):308-319. doi: 10.2337/db24-0890. PMID 39652636